CLINICAL TRIAL: NCT01162369
Title: Validation of Brief Delirium Assessments in Non Critically Ill Hospitalized Patients
Brief Title: Brief Delirium Assessments in Non-Intensive Care Unit (ICU) Patients
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jin H. Han, MD, MSc, Vanderbilt University
Other Study IDs: 100859
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Delirium
Keywords: Delirium, diagnosis, elderly, hospitalization
MeSH Terms: conditions — Delirium; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1 - Non-Delirius Patients
- Group 2 - Delirious Patients

SUMMARY:
Delirium is an acute confusional state characterized by fluctuating mental status, inattention, and either disorganized thinking or an altered level of consciousness. This form of organ dysfunction occurs in up to 50% of hospitalized patients and is associated with worsening mortality, prolonged hospital length of stay, higher health care costs, and accelerated functional and cognitive decline. Despite the negative consequences of delirium, the majority of cases are unrecognized by hospital physicians because it is not routinely screened for. In an effort to facilitate delirium screening, we sought to validate two brief delirium assessments (<2 minutes) in the hospital setting.

DETAILED DESCRIPTION:
Delirium is often missed because physicians do not routinely screen for this diagnosis. Most delirium assessments can take up to 10 minutes to perform making them less likely to be incorporated into the routine physician assessment. Using brief (<2 minutes) and easy to use delirium assessments may ameliorate this quality of care issue. The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) possesses these characteristics, but has only been validated in mechanically and non-mechanically ventilated intensive care unit patients. As a result, it still requires validation in the non-ICU hospitalized patients. Recently, we also developed the Brief Confusion Assessment Method (B-CAM) which is a modification of the CAM-ICU. The benefit is that it takes even less time than the CAM-ICU. However, it also requires validation in hospitalized patients. As result, we propose the following and the following specific aims:

Aim #1: To validate the B-CAM in non-ICU hospitalized patients. The B-CAM will be performed by a clinical trials associate (CTA) and principal investigator in 150 non-ICU hospitalized patients that are > 65 years old. This instrument will be validated against a psychiatrist's Diagnostic and Statistical Manual of Mental Disorders, 4th. Edition Text Revision assessment as the reference standard.

Aim #2: To validate the CAM-ICU in non-ICU hospitalized patients. The CAM-ICU will be performed by a clinical trials associate (CTA) and principal investigator in approximately 150 non-ICU hospitalized patients that are > 65 years old. This instrument will be validated against a psychiatrist's Diagnostic and Statistical Manual of Mental Disorders, 4th. Edition Text Revision assessment as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or greater
* In the non-ICU inpatient setting
* Consulted and evaluated by psychiatry

Exclusion Criteria:

* Severe mental retardation or dementia
* Baseline communication barriers such aphasia, deafness, blindness, or who are unable to speak English
* Refusal of consent
* Previous enrollment
* Comatose
* Out of hospital before the assessments are completed

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The participants will be those who are Vanderbilt University Hospital inpatients aged 65 years or older. There will be no selection bias in regards to race or gender. Only those who meet the inclusion/exclusion criteria will be considered for study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
B-CAM sensitivity and specificity compared with the psychiatrist reference assessment. | day of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jin H Han, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Vanderbilt University Hospital, Nashville, Tennessee
  - Vanderbilt Emergency Medicine, Nashville, Tennessee